CLINICAL TRIAL: NCT06308549
Title: MyDiaMate For Remission Of Diabetes Distress In Type 1 Diabetes (MyREMEDY): A Multi-National Randomised-Controlled Trial
Brief Title: MyDiaMate For Remission Of Diabetes Distress In Type 1 Diabetes (MyREMEDY)
Acronym: MyREMEDY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maartje de Wit (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); King's College London (Other); University of Malaga (Other); Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Responsible Party: Sponsor-Investigator, Maartje de Wit, Principal Investigator, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023.0714
Record Dates: First submitted 2024-02-15; First posted 2024-03-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes; Diabetes Distress
Keywords: Type 1 Diabetes; Diabetes Distress; Self-help; e-health
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 2/3 of participants will be randomised into this arm. They will receive access to MyDiaMate in the language of their participation country for 6 months.
  Interventions: Behavioral: MyDiaMate
- Care As Usual (No Intervention): 1/3 of participants will be randomised into this arm. They will receive Care As Usual, so no intervention, for 3 months. After 3 months, they receive access to MyDiaMate, if so wished.

INTERVENTIONS:
Behavioral: MyDiaMate — MyDiaMate programme
  Arms: Intervention

SUMMARY:
In the MyREMEDY study the investigators research whether the MyDiaMate self-help application is effective in strengthening the mental health of adults with type 1 diabetes in comparison with care as usual. The MyREMEDY study takes place in four countries: The Netherlands, United Kingdom, Spain, and Germany.

DETAILED DESCRIPTION:
Rationale: Type 1 diabetes is a disease that asks constant attention, self-care activities and responsibility from the diagnosed person for the duration of their entire life. Because of this constant burden, many people with type 1 diabetes experience mental health problems such as fatigue, excessive worrying about their blood glucose (especially about dangerously low blood glucose), or eating problems. However, most people with type 1 diabetes who experience such symptoms do not receive professional help. This can have multiple reasons. Oftentimes, the problems are not severe enough to be classified as a disorder. Some people also prefer to work on the problems on their own, at their own pace. For people who experience mental health problems around their diabetes and to support them individually with as little barriers as possible, MyDiaMate was developed.

Objective: To investigate the effectiveness of MyDiaMate in reducing mental health problems in adults with type 1 diabetes who experience distress related to their disease across four countries (NL, DE, UK, ES).

Study design and procedure: Multi-national randomised-controlled trial (intervention : wait-list control group, randomised 2:1 per country).

After screening has confirmed study participation, participants will:

1. Complete the baseline assessment and be randomisation afterwards
2. Use MyDiaMate for 3 months in case of intervention group membership, or get care as usual in case of waitlist control group membership
3. At 3 months, all participants fill in the first follow-up assessment. Additionally, intervention group members will be asked about their satisfaction with and opinion on MyDiaMate (questionnaire and interviews).
4. All participants then receive access to MyDiaMate for the remaining 3 months of the study.
5. At 6 months, all participants complete the second follow-up assessment. Afterwards, the study ends for all participants and access to MyDiaMate is revoked.

Study population: Adults with type 1 diabetes who have been diagnosed more than 6 months ago and who experience distress in relation to their type 1 diabetes.

Intervention: The intervention group receives access to the online self-help programme MyDiaMate for 6 months. MyDiaMate is focused on mental health in type 1 diabetes. It includes psychoeducation and teaches coping strategies that are based on cognitive-behavioural therapy concepts. Moreover, videos in which people with type 1 diabetes talk about their experiences in coping with the disease are embedded in MyDiaMate. MyDiaMate users can also choose to make use of diaries and a module that helps with setting realistic goals. MyDiaMate can be accessed via a private mobile phone, tablet, or laptop/computer whenever wished. Because MyDiaMate is self-help, there is no schedule in when/how much participants should access MyDiaMate. Participants can make use of MyDiaMate as much as they want to, in a way that suits them best personally. Members in the waitlist control group receive access to MyDiaMate after 3 months, for 3 months, if so wished. They too can make use of MyDiaMate in a way that fits their personal time and needs best.

Main study parameters/endpoints: The main study outcome is change in diabetes distress in the intervention group between the baseline and the 3 months assessment. Secondary study outcomes are changes in emotional well-being, psychological self-efficacy in relation to diabetes, social engagement, and fatigue between the baseline and the 3 months assessment in participants from the intervention group. Moreover, in line with the secondary objective, the investigators will make use of MyDiaMate log data such as time spent in MyDiaMate and frequency of use in participants of the intervention group across the first 3 months and investigate in relation to the main and secondary outcomes as well as descriptive data such as age or gender, for which subgroup of MyDiaMate users the application programme is most effective.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no risks related to use of MyDiaMate. The burden of study participation is low, as participants are not instructed to use MyDiaMate in a certain way/intensity and filling in the non-invasive study questionnaires takes around 2 hr in total and is spread across 6 months. Both the intervention and control group have access to MyDiaMate during study participation (for 6 months in case of intervention group membership, for 3 months after 3 months in case of wait-list control group membership). Study participants benefit from study participation because they receive access to MyDiaMate, which may possibly help them with improving the diabetes-related mental health and teaches a variety of type 1 diabetes specific coping strategies, all of which is based on well-researched concepts of psychoeducation and cognitive behavioural therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old at signing the informed consent form
* Type 1 diabetes diagnosis at least 6 months ago
* Having access to the internet and a smartphone/tablet/laptop'/computer for the entire time of study participation
* Experiencing diabetes distress (checked during a phone call between research assistant and participant. The condition is met if the participant has an average score of ≥2 on the 2-item Diabetes Distress Scale (DDS-2), representing clinically meaningful diabetes distress)

Exclusion Criteria:

* Having been diagnosed with a psychiatric disorder in the past 6 months for which the person is under psychological/psychiatric treatment
* Suicidality
* Having started a treatment with psychotropic medication in the past 3 months
* Illiteracy
* Experience of cognitive problems that hamper using MyDiaMate or vision/auditory problems that are hindering in daily life
* Prior use of MyDiaMate (only applicable to participants in the Netherlands)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | Diabetes Distress will be assessed at 0 months (baseline), 3 months (intervention effects), and after 6 months (follow-up).
  Diabetes Distress will be assessed through the 20-item Problem Areas In Diabetes questionnaire (=PAID-20). The Problem Areas In Diabetes questionnaire measures diabetes distress on a 5-point Likert scale ranging from 1 (Not a problem) to 5 (Serious Problem). A higher score represents higher diabetes distress.

SECONDARY OUTCOMES:
Emotional well-being | Emotional well-being will be assessed at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up).
  Emotional well-being will be operationalised as the score on the 5-item World Health Organization Well-Being Index (=WHO-5). The score on the WHO-5 is measured on a 6-point scale ranging from 0 (At no time) to 5 (All of the time) with a lower score representing less emotional well-being.
Psychological self-efficacy in relation to diabetes | Psychological self-efficacy in relation to diabetes will be assessed at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up).
  Operationalised through the Short form of the Diabetes Empowerment Scale (=DES-SF). Psychological self-efficacy in relation to diabetes is assessed on a 5-point scale ranging from 0 (Strongly disagree) to 4 (Strongly agree), with higher scores representing higher psychological self-efficacy in relation to diabetes.
Social Engagement | Social Engagement will be measured at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up)
  Social Engagement will be assessed through the 6-item Lubben Social Network Scale (LSNS-6). The Lubben Social Network Scale measures Social Engagement on a 6-point scale ranging from 0 (None) to 5 (Nine or more). A higher score represents higher social engagement.
Fatigue | Fatigue will be measured at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up)
  Fatigue will be assessed through the 8-item Fatigue subscale of the Checklist Individual Strength (=CIS-F). The Fatigue subscale of the Checklist Individual Strength consists of both positively and negatively framed items that are measured on a 7-point scale ranging from 1 (No, that is not true) to 7 (Yes, that is true). The positively framed items (e.g., I feel fit) will be reverse coded. A higher score will therefore represent stronger fatigue.
HbA1c | Glycaemic control measures, in this case Haemoglobine A1c, will be self-reported at 0 months (baseline), 3 months (intervention effect), and 6 months (follow-up)
  Participants will self-report various outcome measures typical for assesseing glycaemic control in type 1 diabetes. One of these measures is the self-reported Haemoglobine A1c (=HbA1c) value. HbA1c will be measured on different scales, depending on clinical norms of the participating country. This will either be in percentage or mmol/mol. There is no formal minimum or maximum value of HbA1c, although realistically values will be in between 5 and 12 when measured in percentage, or 30 and 100 when measured in mmol/mol. For both scales, a lower score represents better glycaemic control. For data analysis, all scores measured in percentage will be transformed to a HbA1c value measured in mmol/mol.
Time in/above/below range | Glycaemic control measures, in this case time in/above/below range, will be self-reported at 0 months (baseline), 3 months (intervention effect), and 6 months (follow-up)
  Participants will self-report various outcome measures typical for assesseing glycaemic control in type 1 diabetes. One of these measures is the self-reported time in/above/below range. Participants can indicate their own personal target range for blood glucose values, and then indicate the percentage of time during which they were in, above, and below this personal range across the past 14 days. A higher percentage for time in range represents better glycaemic control. A lower percentage for time above range and time below range represents worse glycaemic control.
Events of ketoacidosis/severe hypoglycaemia | Glycaemic control measures, in this case frequency of events of ketoacidosis and severe hypoglycaemia, will be self-reported at 0 months (baseline), 3 months (intervention effect), and 6 months (follow-up)
  Participants will self-report various outcome measures typical for assesseing glycaemic control in type 1 diabetes. One of these measures is the self-reported frequency of events of ketoacidosis and severe hypoglycaemia across the past 12 months when measured at baseline, and across the past 3 months when measured at the 3 and 6 months assessment, respectively. A higher self-reported frequency of events of ketoacidosis and/or severe hypoglycaemia represents worse glycaemic control.

OTHER OUTCOMES:
MyDiaMate usage data | 3 months
  We will passively collect data of MyDiaMate usage through the platform on which MyDiaMate is running (Minddistrict). In practice, we will record the minutes spent in the MyDiaMate application, specifically the minutes spent within each MyDiaMate module, for all members of the intervention group, for 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maartje de Wit, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (4):
- Forschungsinstitut Diabetes-Akademie Bad Mergentheim, Bad Mergentheim, Baden-Wurttemberg, Germany
- Amsterdam UMC, Amsterdam, North Holland, Netherlands
- Universidad de Málaga, Málaga, Spain, Spain
- King's College London, London, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared at reasonable request due to sensitive data.

REFERENCES:
- [Derived] Mohr TC, de Wit M, Embaye J, Ehrmann D, Hermanns N, Lehmann G, Anarte Ortiz MT, Torreblanca Murillo L, Winkley K, Famiglietti A, Pouwer F, Snoek FJ. Effectiveness of the MyDiaMate application in reducing diabetes distress in adults with type 1 diabetes: Study protocol of the multi-national, randomised-controlled MyREMEDY trial. Diabet Med. 2025 Jan;42(1):e15442. doi: 10.1111/dme.15442. Epub 2024 Sep 30. PMID 39350441
- See also: MyREMEDY - Dutch research website — https://myremedyonderzoek.nl/